CLINICAL TRIAL: NCT06903637
Title: Personalized Rehabilitation for Lower Limb Amputation: the Role of Hierarchical Cluster Analysis in Identifying Priority Clinical Variables
Brief Title: Identification of Priority Clinical Variables in Rehabilitation of Lower Extremity Amputation
Acronym: Amputation
Status: Completed | Type: Observational
Sponsor: Cigdem Cinar (Other)
Responsible Party: Sponsor-Investigator, Cigdem Cinar, Associate professor doctor, Biruni University
Organization: Biruni University (Other)
Other Study IDs: 2015-KAEK-80-23-45
Record Dates: First submitted 2025-03-24; First posted 2025-03-31 (Actual); Last update posted 2025-03-31 (Actual); Status verified 2025-03

CONDITIONS: Lower Limb Amputation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Hierarchical Cluster Analysis — The complexity of clinical follow-up stems from the wide range of variables involved, such as physical performance, mobility, pain, psychological well-being, and prosthetic functionality. Therefore, developing methods to identify the most relevant and interrelated clinical variables is critical for enhancing patient management. To address this need, Hierarchical Cluster Analysis (HCA) offers a powerful multivariate statistical approach for detecting relationships among clinical variables.
  Other Names: Houghton Scale; Timed Up and Go Test; rinity Amputation and Prosthesis Experience Scales; 12-item Short Form Health Survey; Locomotor Capabilities Index-5; Medicare Functional Classification Level; Fall Efficacy Scale

SUMMARY:
Background: Identifying which variables influence the personalized rehabilitation of patients with lower limb amputation and understanding their interrelationships optimizes resource allocation. This study aims to identify priority variables that influence clinical follow-up using hierarchical cluster analysis (HCA).

Methods: Data on 26 variables were collected from 70 patients diagnosed with lower limb amputation; (age, gender, body mass index(BMI), marital status, education, occupation, smoking and alcohol use, amputation - level/duration/lateral/etiology, prosthesis type, type of additional prosthesis, Kellgren Lawrence Classification(KLC) - right/left knee, Houghton Scale(HS), Timed-Up&Go(TUG) Test, Trinity Amputation and Prosthesis Experience Scales(TAPES)-prosthesis satisfaction/psychosocial adjustment/activity limitation, Using the 12-item Short Form Health Questionnaire(SF-12)-physical score(PS)/mental score(MS), Locomotor Capabilities Index-5(LCI-5), Medicare Functional Classification Level(MFCL) and Falls Efficacy Scale(FES)). From the collected data, dendrograms were formed by using HCA with Ward linkage method.

ELIGIBILITY:
Inclusion Criteria:

1. having been diagnosis of lower limb amputation,
2. sufficient perceptual acuity to complete the tasks,
3. no head injury within the last 2 years, and
4. being a native Turkish speaker.

Exclusion Criteria:

1. being unable to complete the study,
2. having a history of severe psychiatric illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with lower limb amputation
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2023-12-23 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Houghton Scale | 10 minutes
  This tool categorizes walking ability among lower limb amputees: independent ambulation in the community (score ≥9), independent ambulation in the home or limited community (score 6-8), and limited ambulation in the home (score ≤5)
Timed Up and Go (TUG) Test | 5 minutes
  This test assesses balance and fall risk. Performance categories were as follows: ≤10 seconds (normal mobility), ≤20 seconds (good mobility, can walk without assistance), ≤30 seconds (needs gait aid, cannot walk outside independently). A score of ≥14 seconds indicates a high fall risk
Trinity Amputation and Prosthesis Experience Scales | 10 minutes
  TAPES is a 33-item self-reported questionnaire measuring psychosocial adaptation, activity restriction, and prosthetic satisfaction. The subscales include general adjustment, social adjustment, and adjustment to limitation, along with functional and aesthetic satisfaction
Short-Form Health Survey score | 10 minutes
  (SF-12) is a 12-item, self-rated, health quality instrument and it was validated into many languages as well as for many diseases. It has eight domains represented with one or two questionnaire items; these domains are physical functioning, role participation with physical health problems (role-physical), bodily pain, general health, vitality, social functioning, role participation with emotional health problems (role-emotional), and mental health. It consists of 12 items where two of the items are three-point Likert type, the others are five-point Likert type
The Locomotor Capabilities Index-5 | 10 minutes
  (LCI-5) is a 14-item questionnaire specifically designed to measure walking ability of lower-limb amputees. Two subscales emerge from this general construct; basic abilities (7 items) and advanced abilities (7 items). The items inquire about the ability to perform activities and the level of independence while performing these activities. Each of the 14 items is graded on a 4-point ordinal scale; 0 (not able to), 1 (yes, with help from other person), 2 (yes, with supervision) and 3 (yes, independently). The total LCI score is the sum of the item scores and can range from 0 (worst) to 42 (best). Similarly, subscale scores for basic and advanced capabilities with the prosthesis can range from 0 to 21
Medicare Functional Classification Level | 10 minutes
  (MFCL) is a classification system that categorizes the ambulatory potential of patients with lower limb amputations according to their functional mobility. The classification ranges from K0 (no prosthetic potential) to K4 (high functional potential for advanced physical activities)
Falls Efficacy Scale | 10 minutes
  FES is a test used to assess participants' fear of falling and confidence in performing daily activities without falling. It is a 10-item self-report questionnaire that assesses perceived confidence in performing activities of daily living (e.g. dressing, bathing) without falling. Each item is scored on a 10-point Likert scale; 1 = very confident and 10 = not confident at all, with higher scores indicating greater fear of falling and lower self-efficacy. The total score ranges from 10 to 100

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The following data can be shared as individual participant data. These data were obtained by recording the clinical examination data of the patients in the questionnaire form (does not include personal data such as name, surname, telephone, address)
  ''Houghton Scale, Timed Up and Go Test, Trinity Amputation and Prosthesis Experience Scales (TAPES) - Prosthesis Satisfaction / Psychosocial Adjustment / Activity Restriction, 12-item Short Form Health Survey (SF-12) - Physical Score (PS) / Mental Score (MS), Locomotor Capabilities Index-5 (LCI-5), Medicare Functional Classification Level (K level), and Fall Efficacy Scale.''

REFERENCES:
- [Background] Wade DT. What is rehabilitation? An empirical investigation leading to an evidence-based description. Clin Rehabil. 2020 May;34(5):571-583. doi: 10.1177/0269215520905112. Epub 2020 Feb 10. PMID 32037876